CLINICAL TRIAL: NCT01393457
Title: Cognitive-enhancing DA Medications for Cocaine Dependence
Brief Title: Cognitive Remediation for Cocaine Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Joy Schmitz, Professor - Psychiatry, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DA030787
Record Dates: First submitted 2011-07-11; First posted 2011-07-13 (Estimated); Results first posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Cocaine Dependence
Keywords: cocaine; cognition; medication; treatment
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — carbidopa, levodopa drug combination; ropinirole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ldopa + ropinirole low dose (Active Comparator): levodopa/carbidopa 800/200 mg/d plus ropinirole 2 mg/d
  Interventions: Drug: levodopa/carbidopa; Drug: Ropinirole 2 mg/d
- ldopa + ropinirole high dose (Active Comparator): levodopa/carbidopa 800/200 mg/d plus ropinirole 4 mg/d
  Interventions: Drug: levodopa/carbidopa; Drug: Ropinirole 4 mg/d
- ldopa (Active Comparator): levodopa/carbidopa 800/200 mg/d
  Interventions: Drug: levodopa/carbidopa
- placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: levodopa/carbidopa — 800/200 mg/d
  Other Names: ldopa
  Arms: ldopa; ldopa + ropinirole high dose; ldopa + ropinirole low dose
Drug: Ropinirole 2 mg/d — 2 mg/d
  Other Names: Requip
  Arms: ldopa + ropinirole low dose
Drug: Placebo — sugar pill
  Arms: placebo
Drug: Ropinirole 4 mg/d — 4 mg/d
  Other Names: Requip
  Arms: ldopa + ropinirole high dose

SUMMARY:
The purpose of this study is to evaluate treatments designed to improve cocaine treatment success by combining medications that target cocaine-related cognitive impairments.

ELIGIBILITY:
Inclusion Criteria:

* meet criteria for cocaine dependence
* seeking treatment for cocaine dependence
* be in acceptable health based on medical history and physical exam

Exclusion Criteria:

* dependent on drugs other than cocaine, nicotine, marijuana
* have a medical condition contraindicating treatment with study medications
* having conditions of probation or parole requiring reports of drug use to officers of the court

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 119 (Actual)
Dates: Start 2011-06; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Behavioral and Biomedical Sciences Building, Houston, Texas, United States

REFERENCES:
- [Derived] Suchting R, Green CE, de Dios C, Vincent J, Moeller FG, Lane SD, Schmitz JM. Citalopram for treatment of cocaine use disorder: A Bayesian drop-the-loser randomized clinical trial. Drug Alcohol Depend. 2021 Nov 1;228:109054. doi: 10.1016/j.drugalcdep.2021.109054. Epub 2021 Sep 23. PMID 34600245

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 119 were enrolled (that is, signed the consent); however, only 110 were randomized. Of the 9 that were not enrolled but not randomized, 1 was no longer interested after signing the consent, and 8 were lost to follow up.
Period: Overall Study
Arm/Group | Ldopa + Ropinirole Low Dose | Ldopa + Ropinirole High Dose | Ldopa | Placebo
Started | 26 | 26 | 31 | 27
Completed | 14 | 14 | 16 | 15
Not Completed | 12 | 12 | 15 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ldopa + Ropinirole Low Dose | Ldopa + Ropinirole High Dose | Ldopa | Placebo | Total
Number analyzed (Participants) | 26 | 26 | 31 | 27 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.96 (6.50) | 46.04 (8.70) | 48 (7.87) | 47.11 (8.56) | 46.6 (7.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 5 | 6 | 25
  Male | 19 | 19 | 26 | 21 | 85
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 19 | 19 | 26 | 20 | 84
  White | 2 | 1 | 3 | 3 | 9
  More than one race | 1 | 0 | 0 | 1 | 2
  Unknown or Not Reported | 4 | 6 | 2 | 3 | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 26 | 31 | 27 | 110
Number of days of cocaine use over the last 30 days [Mean (Standard Deviation); unit: days] | 16.12 (8.08) | 16.31 (9.64) | 17.19 (8.46) | 14.74 (8.69) | 16.13 (8.65)

OUTCOME MEASURES:

1. Primary Outcome: Cocaine Use Based on Urine Drug Screening
Description: The mean of the predicted probabilities (derived from generalized linear mixed models) of negative drug screens over all 10 weeks is reported, as per the analysis proposed in the protocol.
Time Frame: 10 weeks
Population: intention to treat
Measure: Mean (Standard Deviation); unit: number of negative drug screens
Arm/Group | Ldopa + Ropinirole Low Dose | Ldopa + Ropinirole High Dose | Ldopa | Placebo
Number analyzed (Participants) | 26 | 26 | 31 | 27
number of negative drug screens | 20.36 (29.51) | 15.57 (21.96) | 22.3 (28) | 27.8 (30.35)

2. Secondary Outcome: Number of Participants Who Completed the 10 Week Trial
Time Frame: 10 weeks
Measure: Number; unit: participants
Arm/Group | Ldopa + Ropinirole Low Dose | Ldopa + Ropinirole High Dose | Ldopa | Placebo
Number analyzed (Participants) | 26 | 26 | 31 | 27
participants | 14 | 14 | 16 | 15

ADVERSE EVENTS:
Time Frame: weekly for 10 weeks
Description: Side effects were not considered to be adverse events.
Arm/Group | Ldopa + Ropinirole Low Dose | Ldopa + Ropinirole High Dose | Ldopa | Placebo
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26 | 0/31 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/26 | 1/26 | 0/31 | 3/27
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/31 | 0/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ldopa + Ropinirole Low Dose (N=26) | Ldopa + Ropinirole High Dose (N=26) | Ldopa (N=31) | Placebo (N=27)
Chest pain (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight gain (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gout flare up (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicide ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2011-09-02): https://cdn.clinicaltrials.gov/large-docs/57/NCT01393457/Prot_000.pdf
  • Statistical Analysis Plan (2011-09-02): https://cdn.clinicaltrials.gov/large-docs/57/NCT01393457/SAP_001.pdf